CLINICAL TRIAL: NCT04906603
Title: Theta Burst Stimulation for Headaches After Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Minnesota Office of Higher Education (Other Government); The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cristina Sophia Albott, Physician, Minneapolis Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAM-19-00458
Record Dates: First submitted 2021-05-04; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Post-Traumatic Headache; Transcranial Magnetic Stimulation; Brain Injuries, Traumatic; Quality of Life
MeSH Terms: conditions — Post-Traumatic Headache; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TBS Headache (Experimental)
  Interventions: Device: Theta Burst Stimulation

INTERVENTIONS:
Device: Theta Burst Stimulation — TBS will be administered three times per day and three days per week for four weeks (totaling 12 TBS intervention visits and 36 TBS intervention sessions). Each TBS intervention session will last approximately 10 minutes (stimulation parameters = 50 Hz, 3 pulses, 10 bursts, 10 second cycle time, 60 cycles, 1800 total pulses).

SUMMARY:
The purpose of this study is to evaluate if theta burst stimulation (TBS) can reduce chronic headaches caused by a traumatic brain injury (TBI). TBS is a safe, drug-free brain stimulation technique that uses magnets to create electricity and stimulate nerve cells in the brain. After repeated TBS sessions, the increased stimulation of nerve cells can alter the way the brain communicates with itself (by creating new neural pathways) which, in turn, can reduce pain symptoms. Participants in this study will complete a baseline assessment followed by four weeks of daily home headache assessment. Participants will then receive four weeks of TBS administered three times per day and three days per week. After TBS is completed, participants will complete an additional four weeks of daily home headache assessment and return for a one-month follow-up assessment. Participation is expected to last three months.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the safety and efficacy of theta burst stimulation (TBS) for the management of post-traumatic headaches to improve outcomes and quality of life for individuals who have suffered a traumatic brain injury (TBI). To improve tolerability and logistical burden, we have developed a novel design whereby participants will receive three doses of TBS on alternate days of the week. This design will allow us to assess efficacy while leveraging an accelerated treatment course (nine stimulation sessions per week). We have three specific aims:

Specific Aim 1. To determine the efficacy and safety of TBS for the treatment of post-traumatic headache among individuals who have sustained a mild TBI. Hypothesis 1a: TBS will be safe, well-tolerated, and reduce the number of headache days. Hypothesis 1b: TBS will improve function and quality of life outcomes.

Specific Aim 2: To determine the efficacy and safety of an accelerated time-course of TBS for the management of post-traumatic headache. Hypothesis 2a: The accelerated-time course will be safe, well-tolerated, and improve quality of life outcomes. Hypothesis 2b: The accelerated time-course will produce greater and faster improvement in headache symptoms than that reported in the literature for standard repetitive transcranial magnetic stimulation (rTMS) protocols.

Specific Aim 3: To examine the durability of treatment response to accelerated TBS during a one-month observational period. Hypothesis 3: Accelerated TBS will result in enduring treatment response of post-traumatic headache symptoms over the follow-up period.

This study will be an open-label pilot study and will enroll 20. Participants will complete four weeks of pre-intervention headache assessment via Ecological Momentary Assessment (EMA). Participants will then receive TBS intervention three times a week for four weeks. TBS will be administered in 10-minute sessions, three times per day with 20 minutes between sessions. TBS intervention will be completed using the Magstim Horizon Performance Transcranial Magnetic Stimulation (Magstim Company, Ltd.) device or the MagVenture MagPro X100 with MagOption Transcranial Magnetic Stimulation device (MagVenture, Inc.). Both devices are FDA-cleared to provide TBS for the treatment of Major Depressive Disorder and will be used off-label for this study. After TBS intervention, participants will complete an additional four weeks of EMA headache assessment and return for a one-month follow-up assessment. Participants will be assessed with multiple instruments and at multiple timepoints including interviews, questionnaires, and cognitive functioning assessments.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving services through the MVAHCS
* History of mild TBI according to VA/DoD Clinical Practice Guidelines (2009) with one or more of the following criteria present after head injury:

  * Loss of consciousness between 0-30 minutes
  * Post-traumatic amnesia between 0-24 hours
  * Alteration of consciousness/mental state up to 24 hours
  * Glasgow Coma Score between 13-15 (best available score within first 24 hours)
* Post-traumatic headaches defined by International Classification for Headache Diagnosis 3rd Edition (ICHD-3) guidelines with the following criteria present:

  * Headaches developing within seven days following trauma or injury to the head and/or neck
  * Headaches persisting beyond three months
* Chronic daily headaches defined by clinical standards with the following criterion present:

  o 15 or more headache days per month
* Men and women 18-75 years of age
* Possess a smartphone and agree to download and use the EMA application on their personal device
* Capable and willing to provide voluntary informed consent

Exclusion Criteria:

* History of moderate or severe TBI according to VA/DoD Clinical Practice Guidelines (2009) with one or more of the following criteria present after head injury:

  * Loss of consciousness greater than 30 minutes
  * Post-traumatic amnesia greater than 24 hours
  * Worst Glasgow Coma Scale less than 13 within the first 24 hours unless invalidated upon review (e.g., attributable to intoxication, sedation, systemic shock)
  * Abnormal structural imaging
* Current (within six months of enrollment) psychosis and mania
* Current (within one month of enrollment) substance dependence with the exclusion of opioids
* Personal history of epilepsy or seizure disorder

  o Does not include seizures therapeutically-induced by ECT or identified as a single seizure event (based on the principal investigator's judgement)
* Metal particles in the eye or head (exclusive of the mouth) (e.g., shrapnel, fragments from welding or metalwork, etc.)
* Implanted medical device above the clavicle (e.g., aneurysm clips, shunts, stimulators, cochlear implants, electrodes, etc.)
* Significant neurological disorder or insult that would impact risk (based on the principal investigator's judgement and research literature)
* Current use of medications with significant potential for lowering seizure threshold
* Current benzodiazepine usage at a dose higher than 3mg of lorazepam or equivalent
* Electroconvulsive therapy (ECT) or cortical energy exposure within one month of enrollment (including participation in any other neuromodulation treatments or studies)
* Current (within one month of enrollment) participation in another interventional study that would impact the results of this research
* Inadequate communication (e.g., language barrier)
* Women who are pregnant, trying to become pregnant, or breastfeeding
* Women of childbearing age/potential who are not using a medically-accepted form of contraception when sexually active

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Ecological Momentary Assessment (EMA) for Headache Frequency, Intensity, and Impairment | Participants will take the daily headache assessment every day for 2 weeks pre-intervention, every day for 4 weeks during intervention, and every day for 4 weeks post-intervention to track their change in headache frequency, intensity, and impairment.
  EMA will be used for repeated real-time sampling of headaches symptoms prior to intervention, during intervention, and after intervention. Participants will access the EMA application (app) on their personal smartphones.
World Health Organization Quality of Life Scale (WHOQOL-BREF) | Baseline visit, pre-intervention (2 weeks after baseline), post-intervention (4 weeks after pre-intervention), and at follow-up (1 month post-intervention).
  The WHOQOL-BREF is a 26-item self-report assessment of quality of life and will be used to assess changes in QOL over the course of the study. Items are rated on a scale from 1 (very poor) to 5 (very good).
Migraine Disability Assessment (MIDAS) | Baseline visit, pre-intervention (2 weeks after baseline), post-intervention (4 weeks after pre-intervention), and at follow-up (1 month post-intervention).
  The MIDAS is a 5-item self-report assessment of headache disability and will be used to assess change in headache impairment over the course of the study. Participants are to respond with the number of days they have experienced various types of headache disability. The last question asks them to rate on a scale from 0 (no pain at all) to 10 (pain as bad as it can be).
Patient-Reported Outcomes Measurement Information System - Pain Interference - Short Form 6b (PROMIS-SF6b) | Baseline visit, pre-intervention (2 weeks after baseline), post-intervention (4 weeks after pre-intervention), and at follow-up (1 month post-intervention).
  The PROMIS-SF6b is a 6-item self-report assessment of pain interference and will be used to assess change in universal (non-headache specific) pain over the course of the study. Items are rated on a 5 point scale from "Not at all" to "Very Much".

SECONDARY OUTCOMES:
Barratt Impulsiveness Scale - Version 11 (BIS-11) | Baseline visit, pre-intervention (2 weeks after baseline), post-intervention (4 weeks after pre-intervention), and at follow-up (1 month post-intervention).
  The BIS-11 is a 30-item self-report measure of impulsivity and will be used to assess change in impulsive behavior over the course of the study. Items are rated on a 4 point scale from "Rarely or never" to "Almost always or always".
Beck Anxiety Inventory (BAI) | Baseline visit, pre-intervention (2 weeks after baseline), post-intervention (4 weeks after pre-intervention), and at follow-up (1 month post-intervention).
  The BAI is a 21-item self report assessment of anxiety severity and will be used to assess change in mood over the course of the study. Items are rated on a 4 point scale from "Not at all" to "Severely---it bothered me a lot."
Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR) | Baseline visit, pre-intervention (2 weeks after baseline), post-intervention (4 weeks after pre-intervention), and at follow-up (1 month post-intervention).
  The QIDS-SR is a 16-item self-report assessment of depression severity and will be used to assess change in mood over the course of the study. Each item has 4 choices that specifically tie in to the question. For example:
  Question 1. Falling asleep
  1. I never take longer than 30 minutes to fall asleep
  2. I take at least 30 minutes to fall asleep, less than half the time.
  3. I take at least 30 minutes to fall asleep, more than half the time.
  4. I take more than 60 minutes to fall asleep, more than half the time.
PTSD Checklist for DSM-V (PCL-5) | Baseline visit, pre-intervention (2 weeks after baseline), post-intervention (4 weeks after pre-intervention), and at follow-up (1 month post-intervention).
  The PCL-5 is a 20-item self-report measure of post-traumatic stress disorder (PTSD) symptoms and severity and will be used to assess change in mood over the course of the study. Items are rated on a 5 point scale from "Not at all" to "Extremely".
Dot Counting (Cognitive Task) | The dot counting task will be administered at every stimulation visit during the 4 weeks of intervention (total of 12 times).
  The Dot Counting Task is a computerized measure of verbal working memory.
N-Back (Cognitive Task) | The N-Back task will be administered at every stimulation visit during the 4 weeks of intervention (a total of 12 times).
  The N-Back Task is a continuous performance test that is used to measure working memory and processing speed.
Risk Task (Cognitive Task) | The risk task will be administered at every stimulation visit during the 4 weeks of intervention ( a total of 12 times).
  The Risk Task is a computerized behavioral measure of the propensity for risk taking within a decision making task.
Caffeine and Nicotine Use Questionnaire | Baseline and daily for 10 weeks after baseline
  The Caffeine and Nicotine Use Questionnaire is a proprietary measure used to record typical patterns of caffeine and nicotine use at study baseline. Daily caffeine and nicotine use will then be tracked over the course of the study using EMA.

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Final data sets may be made available upon written request and subject to sponsor approval.